CLINICAL TRIAL: NCT05307419
Title: Prospective Randomised Blinded Study Comparing Full Thickness Biopsy and Rectal Suction Biopsies in the Diagnosis of Mb: Hirschsprung
Brief Title: Full Thickness vs. Rectal Suction Biopsy in the Diagnosis of Hirschsprungs Disease
Acronym: BIOPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S-20190116
Record Dates: First submitted 2022-02-02; First posted 2022-04-01 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprungs disease; Rectal biopsy; Rectal suction biopsy; Full thickness biopsy; Randomised; Blinded; Mb. Hirschsprung
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Intervention Model Description: Prospective randomized blinded case-control study.
Who Masked: Outcomes Assessor
Masking Description: The pathologist is masked by 30 day delay and should be conducted by another pathologist than the first.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectal suction biopsy first (Active Comparator): Children randomised for pahtological evaluation of rectal suction biopsy tissue first.
  Interventions: Procedure: Rectal suction biopsy.; Procedure: Full-thickness rectal biopsy.
- Full thickness biopsy first (Active Comparator): Children randomised for pathological evaluation of full thickness biopsy tissue first.
  Interventions: Procedure: Rectal suction biopsy.; Procedure: Full-thickness rectal biopsy.

INTERVENTIONS:
Procedure: Rectal suction biopsy. — Suction biopsy performed
Procedure: Full-thickness rectal biopsy. — Full-thickness biopsy performed

SUMMARY:
The objective of this prospective study is to compare the diagnostic accuracy of rectal suction biopsy (RSB) compared to full thickness rectal biopsy (FTB) in the diagnosis of Hirschsprungs Disease (HD) in children. The secondary objective to compare cost-effectiveness of the two procedures

DETAILED DESCRIPTION:
Diagnostic procedures involving the need of surgically obtaining tissue material, carry the risk of complications and the risk of being inconclusive due to various reasons. Lowering the risk of inconclusive diagnostic tests with highest sensitivity and specificity is of high importance in all diagnostic procedures.

A full thickness rectal biopsy (FTB) includes both the submucosal and the myenteric nerve plexus for histological evaluation for presence of ganglion cells and hypertrophic nerve fibers. FTB is performed in general anesthesia (GA), the biopsy is cut with scissors under direct visualization of the intestine and with suturing of the biopsy defect. The other method is a suction biopsy (RSB) in which the biopsy is more superficial acquiring only the submucosal layers. RSB's are performed with a specially designed rectoscope, and the biopsy is obtained under negative pressure within the scope, without visual guidance. This procedure can be performed without anesthesia in children blow 1 year and does not necessitate suturing of the bowel.

The problem with especially RSB could be that the biopsy is too superficial or too small in size for proper pathological evaluation. As a consequence the child has to undergo a new procedure. There is also the risk of false positive or false negative results, which is a serious clinical issue carrying the risk of performing extensive surgery in an otherwise healthy child.

Inconclusive biopsies differ extensively from series to series. But the two largest studies show a rate of inconclusive biopsies at 10% for RSB and 5% for FTB.(Freidmacher and Bjorn). The biopsy profile is similar with less than 1% severe complications (Above Clavien DindoIII) in both procedures, with bleeding as dominating in RSB and Fever in FTB.

Thus there are different advantages and disadvantages between the two methods of biopsy in children suspicious of HD, and different centers advocate either. A prospective comparison of both methods with the child as its own control is a more precise way to compare the two methods and has never been performed. Thus, this study is expected to give an answer to an important research question that will have potential implication worldwide.

Hypothesis:

Our hypothesis is that FTB has lower rate of inconclusive biopsies compared to RSB in the diagnosis of HD.

Design:

Prospective, biopsy sample randomised study.

Method:

Patients referred for rectal biopsy at Odense University Hospital on the suspicion of HD will undergo both an FTB and RSB performed under GA in the same procedure.

Patients will be randomised to which biopsy will be examined first at the pathology department. If a diagnosis can bed securely made on the first tissue samples the other biopsy materials will be stores for examination by another pathologist 30 days later. If any nerve cell is present the sample is negative for Mb. Hirschsprung. If no nervecells is present the biopsy the patient is positive for mb. Hirschsprung. If the tissue is evaluated as not suitable for diagnosis the sample is inconclusive. If the sample is inconclusive the tissue from the other biopsy method is evaluated immediately to secure a fast diagnosis.

All children between 0-15 years of age undergoing biopsies for diagnosis of the diagnosis of HD in Western Denmark from 1/9 2020 will be offered to participate and parental accept will be acquired.

Cost-effectiveness will be measured upon with data from pathology cost and surgery utensils cost.

These will be compared between the two groups.

Power calculation:

With the assumption of a 5 % inconclusive rate for FTB and 10% for RSB (2,5) a McNemar's test for matched comparison of dichotomous outcome (inconclusive / conclusive) indicates the need for 282 patients to obtain 70% strength and a significance level of 5%. (P-value 0.05).

These calculations are based on the largest numbers of biopsy evaluations in the literature.

In these publications a rate of 5% inconclusive biopsies at FTB and 10% at RSB are found.

Interim analyse will be performed after 25%, 50% and 75%. Above 8% complications on 30-day follow-up will result in the study will be paused and examinations of the complications will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are referred for rectal biopsy for suspected HD, age 0-15 years.
* Written informed consent of the parents or guardian.

Exclusion Criteria:

* Lack of consent from parents or guardians.
* Previous surgery on the ano-rectum e.g. crohns disease and/or fistulas

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of inconclusive biopsies between FTB and RSB. | 30 days
  Prospective comparison of RSB and FTB when performed on the same patient. Evaluation of diagnostic accuracy.

SECONDARY OUTCOMES:
Surgical and pathology cost. | 30 days
  Cost-effectiveness will be measured from surgical and pathology procedural and utensils costs in euros, between RSB and FTB.

CONTACTS AND LOCATIONS:
Overall Officials: Mark mr Ellebaek, Dr, Study Director — University of Southern Denmark; Rasmus mr Nielsen, Dr, Study Chair — Odense University Hospital; Gunvor ms Madsen, Dr, Study Chair — Odense University Hospital; Niels mr Bjorn, Dr, Principal Investigator — Odense University Hospital; Lene ms Christensen, Dr, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muise ED, Hardee S, Morotti RA, Cowles RA. A comparison of suction and full-thickness rectal biopsy in children. J Surg Res. 2016 Mar;201(1):149-55. doi: 10.1016/j.jss.2015.10.031. Epub 2015 Oct 28. PMID 26850196
- [Background] Bjorn N, Rasmussen L, Qvist N, Detlefsen S, Ellebaek MB. Full-thickness rectal biopsy in children suspicious for Hirschsprung's disease is safe and yields a low number of insufficient biopsies. J Pediatr Surg. 2018 Oct;53(10):1942-1944. doi: 10.1016/j.jpedsurg.2018.01.005. Epub 2018 Jan 31. PMID 29426767
- [Background] Alizai NK, Batcup G, Dixon MF, Stringer MD. Rectal biopsy for Hirschsprung's disease: what is the optimum method? Pediatr Surg Int. 1998 Mar;13(2-3):121-4. doi: 10.1007/s003830050264. PMID 9563023
- [Background] Stewart CL, Kulungowski AM, Tong S, Langer JC, Soden J, Somme S. Rectal biopsies for Hirschsprung disease: Patient characteristics by diagnosis and attending specialty. J Pediatr Surg. 2016 Apr;51(4):573-6. doi: 10.1016/j.jpedsurg.2015.10.047. Epub 2015 Oct 19. PMID 26592956
- [Background] Friedmacher F, Puri P. Rectal suction biopsy for the diagnosis of Hirschsprung's disease: a systematic review of diagnostic accuracy and complications. Pediatr Surg Int. 2015 Sep;31(9):821-30. doi: 10.1007/s00383-015-3742-8. Epub 2015 Jul 9. PMID 26156878
- [Background] Imaizumi T, Murakami H, Nakamura H, Seo S, Koga H, Miyano G, Okawada M, Doi T, Lane GJ, Okazaki T, Arakawa A, Yao T, Yamataka A. Rectal mucosal/submucosal biopsy under general anesthesia ensures optimum diagnosis of bowel motility disorders. Pediatr Surg Int. 2016 Dec;32(12):1173-1176. doi: 10.1007/s00383-016-3976-0. Epub 2016 Sep 23. PMID 27663688
- [Background] Pini-Prato A, Martucciello G, Jasonni V. Rectal suction biopsy in the diagnosis of intestinal dysganglionoses: 5-year experience with Solo-RBT in 389 patients. J Pediatr Surg. 2006 Jun;41(6):1043-8. doi: 10.1016/j.jpedsurg.2006.01.070. PMID 16769331
- [Background] Ali AE, Morecroft JA, Bowen JC, Bruce J, Morabito A. Wall or machine suction rectal biopsy for Hirschsprung's disease: a simple modified technique can improve the adequacy of biopsy. Pediatr Surg Int. 2006 Aug;22(8):681-2. doi: 10.1007/s00383-006-1714-8. Epub 2006 Jul 4. PMID 16821022
- [Background] Hall NJ, Kufeji D, Keshtgar A. Out with the old and in with the new: a comparison of rectal suction biopsies with traditional and modern biopsy forceps. J Pediatr Surg. 2009 Feb;44(2):395-8. doi: 10.1016/j.jpedsurg.2008.10.093. PMID 19231542
- [Background] De Lorijn F, Reitsma JB, Voskuijl WP, Aronson DC, Ten Kate FJ, Smets AM, Taminiau JA, Benninga MA. Diagnosis of Hirschsprung's disease: a prospective, comparative accuracy study of common tests. J Pediatr. 2005 Jun;146(6):787-92. doi: 10.1016/j.jpeds.2005.01.044. PMID 15973319